CLINICAL TRIAL: NCT07088445
Title: Therapeutic Prospects of Faricimab Injection for Patients Affected by Neovascular Age-Related Macular Degeneration
Status: Not yet recruiting | Type: Observational
Sponsor: Hui Peng (Other)
Responsible Party: Sponsor-Investigator, Hui Peng, Chief physician, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2025-155-04
Record Dates: First submitted 2025-06-26; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Neovascular Age-related Macular Degeneration(nAMD)
MeSH Terms: interventions — faricimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Faricimab — Intravitreal injection of 6mg famotizumab into the vitreous cavity of patients with non primary wet age-related macular degeneration

SUMMARY:
Neovascular Age-Related Macular Degeneration (nAMD) is one of the main causes of irreversible vision loss in the elderly, characterized by neovascularization and vascular leakage in the macular area, ultimately leading to damage to retinal structure and visual impairment. At present, anti vascular endothelial growth factor (VEGF) therapy is the main approach for treating nAMD, including VEGF inhibitors such as Aflibercept and Conbercept. However, some patients show decreased treatment tolerance or efficacy after long-term use of these drugs . Faricimab, a bispecific antibody that targets both VEGF and angiopoietin-2 (Ang-2), is expected to provide a new treatment option for patients resistant to existing VEGF therapies due to its unique dual mechanism of action The aim of this study is to explore the treatment response rate and prognosis of farnesyl monoclonal antibody in patients with refractory nAMD, including visual improvement and imaging changes, in order to provide more scientific treatment decision-making basis for clinical practice. At the same time, to determine its efficacy and safety in actual clinical treatment, in order to provide more flexible and personalized treatment options for nAMD patients, reduce their treatment burden, improve treatment compliance and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of wet age-related macular degeneration (nAMD) in individuals aged 50 years to 80 years.
* Refractory nAMD: ≥ 6 injections of anti VEGF drugs within 12 months or ≥ 4 injections within 6 months, CFT ≥300 μm， In addition, there is retinal fluid.
* BCVA is 24 to 73 letters (equivalent to Snellen vision of about 20/40 to 20/320) in the early treatment of diabetes retinopathy study (ETDRS) scoring scale.
* The subjects can understand the purpose of the study and voluntarily sign a written informed consent.

Exclusion Criteria:

* Accompanied by other eye diseases that may affect the structure or function of the macula (such as diabetes retinopathy, uveitis, etc.). There are obvious scars or fibrosis on the vitreous or retina.
* There is uncontrolled hypertension, diabetes or other systemic diseases that may affect the treatment effect.
* Having undergone eye surgery (such as retinal laser treatment or vitrectomy) and less than 3 months after surgery.
* Allergic to farnesyl monoclonal antibody or its components.
* Patients who are unable to complete follow-up or have poor compliance.
* Researchers determine other factors that may affect the safety or data integrity of the experiment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolls patients aged 50-80 years with refractory neovascular age-related macular degeneration (nAMD), defined as persistent disease activity (central subfield thickness ≥300 μm + intra-/subretinal fluid) despite ≥6 anti-VEGF injections within 12 months or ≥4 injections within 6 months. Eligible participants must have a baseline BCVA of 24-73 ETDRS letters (Snellen ~20/40-20/320) and no confounding ocular comorbidities (e.g., diabetic retinopathy, macular fibrosis) or uncontrolled systemic conditions (e.g., hypertension, diabetes). Exclusions include recent ocular surgery (<3 months), drug hypersensitivity, or inability to comply with follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants With a Valid vs. Invalid Response at Month 6 | Month 6
  ① Valid response: a. Good response: No IRF, SRF, and ≥75% reduction in CMT; b. Partial response: Persistent IRF/SRF with a 25-75% reduction in CMT. ② Invalid response: a. Poor response: Persistent or new IRF/SRF with a 0-25% reduction in CMT; b. No response: IRF, SRF, and/or PED remain unchanged or increased.

SECONDARY OUTCOMES:
Change in Best-Corrected Visual Acuity (BCVA) From Baseline | Baseline Month 3 Month 6
  Change in BCVA as measured by ETDRS letter score.
Change in Central Macular Thickness (CMT) From Baseline | Baseline Month 3 Month 6
  Change in central macular thickness measured via OCT
Change in NEI VFQ-25 Score From Baseline | Baseline Month 3 Month 6
  Change in patient-reported visual function based on the NEI VFQ-25 (scale 0-100)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to concerns regarding patient privacy, the limited scope of data use consent obtained from participants, and institutional policies restricting public data disclosure. Additionally, the current study does not have the infrastructure in place to support secure data sharing and oversight.